CLINICAL TRIAL: NCT06623344
Title: Brain Volume and Cardiac Function in Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Canon Medical Systems, USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00418683
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
Keywords: Heart Failure; Cardiovascular Magnetic Resonance Imaging; brain
MeSH Terms: conditions — Heart Failure | interventions — Magnetic Resonance Spectroscopy; Contrast Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospitalized (Other): Participants who were hospitalized due to heart failure (HF) illness.
  Interventions: Other: Magnetic Resonance Imaging with or without Contrast
- Non-Hospitalized (Other): Participants who had heart failure (HF) but did not require hospitalization secondary to the illness.
  Interventions: Other: Magnetic Resonance Imaging with or without Contrast

INTERVENTIONS:
Other: Magnetic Resonance Imaging with or without Contrast — Completion of Magnetic Resonance Imaging of the brain, heart, lungs, and liver with and without contrast.

SUMMARY:
Patients with heart failure (HF) exhibit greater structural brain alterations and higher dementia risks than the general population. Neural atrophy in nearly every region of medical limbic circuit has been observed in HF patients. Reduction of cerebral blood flow has been suggested as the pathophysiological pathway linking HF and structural brain changes. Indeed, lower cardiac index levels were related to lower cerebral blood flow in older adults without stroke, dementia, or heart failure. A few prior studies have examined the subcortical structural differences in patients with HF compared to controls. Brain volume loss (including putamen and hippocampal volumes) have been reported in patients with low ejection fraction. Significant gray matter loss was found in specific brain regions of HF patients and included structures that serve demonstrated roles in cognitive functions. In the investigator's previous study (Comprehensive Imaging Exam of Convalesced COVID-19 Patients - COVID-19 RELATED SUBMISSION-IRB00252436), involving 100 participants (volunteers with normal heart function (ejection fraction; 50%)), the investigators observed significant correlations between thalamic volumes and ventricular stroke volumes in volunteers. Building on these findings, the investigators intend to expand the research to include individuals with heart failure (HF), employing the same MRI protocol. The study will involve obtaining a set of T1-weighted brain images to measure the volumes of seven subcortical structures. The investigators goal is to explore the relationship between subcortical volumes and cardiac parameters. Additionally, the investigators will examine whether patients with HF experience a more rapid reduction in subcortical volumes compared to those with normal cardiac function (EF;50%).

DETAILED DESCRIPTION:
Heart failure (HF) is a multifaceted clinical syndrome characterized by the heart's inability to effectively pump blood to meet the body's demands. This condition often results from various structural or functional cardiac disorders, impacting not only the heart but also multiple organ systems, including the brain, kidneys, lungs, and circulatory system. Patients with heart failure present a spectrum of symptoms that significantly affect quality of life, such as dyspnea and fatigue, and are typically identified by cardiac dysfunction markers like abnormal left or right ventricular filling and elevated filling pressures. Recent advances in diagnostic technologies, particularly in imaging modalities like Cardiovascular Magnetic Resonance Imaging (CMR), have opened new avenues for in-depth exploration of heart failure's underlying pathophysiology. CMR is increasingly used in heart failure management for risk stratification, viability assessment, and diagnosing conditions like myocarditis and cardiomyopathy. This technology enables detailed assessment of myocardial function, structural changes, and interactions with other organ systems. Patients with heart failure exhibit greater structural brain alterations and higher dementia risks than the general population. Neural atrophy in nearly every region of medical limbic circuit has been observed in HF patients. Initial research showed a strong correlation between thalamic volumes and ventricular stroke volumes in healthy volunteers. The investigators plan to extend this study to heart failure (HF) patients using the same MRI methods to assess the connection between subcortical brain volumes and heart health. Additionally, the investigators will explore if HF patients experience a faster decline in these brain volumes than individuals with normal heart function.

- Objectives:

Primary: To access the correlation of cardiac structure and function to the subcortical volumes in patients with heart failure.

Secondary: To compare the correlation between cardiac structure and function and subcortical volumes in heart failure patients with that in participants with normal heart function.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with an ejection fraction (EF) below 50% who are willing to
* provide informed consent.
* Not claustrophobia.
* Age: 21 years and above.
* Ambulatory patients are eligible.

Exclusion Criteria:

* Known allergy to gadolinium contrast agents
* Metal fragments in eyes, brain, or spinal cord
* Glomerular filtration rate (GFR) 45 mL/min (using the Cockcroft-Gault formula)
* Pregnancy
* Internal electrical devices, such as cochlear implant, spinal cord stimulator, pacemaker, or defibrillator
* Presence of any other history or condition that the investigator feels would be problematic
* Severe claustrophobia
* Weight exceeding 300 lbs. (MRI table weight restrictions)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Subcortical Volumes in Heart Failure | From enrollment up to 30 days post treatment
  To access the correlation of cardiac structure and function to the subcortical volumes in patients with heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Joao AC Lima, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Center for Advanced Imaging and Research Science, Johns Hopkins Science + Technology Park at 1812 Ashland Avenue, Baltimore, MD, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may provided to qualified researchers with academic interest in COVID-19. Data shared will not contain any personal health information (PHI). A statement of work and data use agreement are pre-requisites for data sharing.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 12 months after article publication. Data will be made accessible up to 24 months with extensions considered as needed.
Access Criteria: Access provided upon request.